CLINICAL TRIAL: NCT03784430
Title: Soft and Hard Tissue Changes After Immediate Single-tooth Replacement With or Without a Submarginal Connective Tissue Graft
Brief Title: Soft and Hard Tissue Changes After Immediate Single-tooth Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Massimo de Sanctis, Prof., Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Winsix 1
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Implant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implant (Active Comparator): Immediate dental implant placement
  Interventions: Procedure: Immediate dental implant placement
- Implant+CTG (Experimental): Immediate dental implant placement with CTG.
  Interventions: Procedure: Immediate dental implant placement with CTG

INTERVENTIONS:
Procedure: Immediate dental implant placement — Tooth will be extracted and a dental implant will be positioned at the same time.
  Arms: Implant
Procedure: Immediate dental implant placement with CTG — Tooth will be extracted and a dental implant will be positioned at the same time with a connective tissue graft.
  Arms: Implant+CTG

SUMMARY:
A recent systematic review (Lee et al, 2016) reported that placement of a soft tissue graft concurrent with immediate implantation may contribute to the stability of gingival level and the augmentation of soft tissue contour. However, most included studies did not have a control group to directly demonstrate the benefit of an immediate implant combined with soft tissue graft (IMITG) compared to immediate implant alone.The objective of this randomized controlled clinical trial with a parallel design is to evaluate the influence of the connective tissue graft on the buccal bone alterations after tooth extraction and immediate implant placement by means of cone beam computer tomography (CBCT).

DETAILED DESCRIPTION:
All participants will be selected on a consecutive basis, among individuals, above the age of 18 years, referred to Dental Clinic of the San Raffaele University, with a single failing tooth in the upper and lower jaw from second premolar to second premolar, candidates for a single implant restoration. After local anesthesia, a split-full-split thickness envelope flap, as described for the treatment of multiple gingival recessions by Zucchelli and de Sanctis (2000), will be elevated and the tooth will be extracted a-traumatically. The immediate implantation procedure will be carried out according to the manufacture protocol and 1mm of the transmucosal portion of the implant will be positioned under the buccal bone crest. In the group "Implant+CTG" a connective tissue graft (CTG), resulting from the extraoral de-epithelialization with the knife blade of a free gingival graft harvested from the palate, will be anchored at the anatomic papillae with 2 horizontal mattress sutures and positioned 1 mm coronal to the buccal bone crest and in the apical direction 2 mm above the buccal crest. Patients will be followed for 6 months after implant placement and 6 months after loading.

ELIGIBILITY:
Inclusion Criteria:

* a single tooth to be extracted for endodontic failure, fractures, root caries or resorption in the maxillary and mandibular area from second premolar to second premolar
* patient in good systemic health, with no contraindication for oral surgical interventions

Exclusion Criteria:

* patients with impaired systemic diseases that will interfere with surgical interventions (autoimmune diseases, uncontrolled diabetes)
* assumption of bisphosphonate
* smoking more than 10 cigarettes a day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Volumetric buccal bone changes | 6 months
  Ratio scale - lower values represent a better outcome

SECONDARY OUTCOMES:
Volumetric buccal soft tissue changes | 6 months
  Ratio scale - higher values represent a better outcome
Buccal soft tissue changes | 6 months
  Ratio scale - higher values represent a better outcome
Patient perception outcomes | 1 week and 6 months
  Visual Analogic Scale - values from '0=no pain' to '10=worst pain imaginable'

CONTACTS AND LOCATIONS:
Overall Officials: Massimo de Sanctis, MD, Principal Investigator — Università Vita-Salute San Raffaele
Locations (1):
- Massimo de Sanctis, Milan, Mi, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schneider D, Schmidlin PR, Philipp A, Annen BM, Ronay V, Hammerle CH, Attin T, Jung RE. Labial soft tissue volume evaluation of different techniques for ridge preservation after tooth extraction: a randomized controlled clinical trial. J Clin Periodontol. 2014 Jun;41(6):612-7. doi: 10.1111/jcpe.12246. Epub 2014 Mar 26. PMID 24593810
- [Background] Jung RE, Philipp A, Annen BM, Signorelli L, Thoma DS, Hammerle CH, Attin T, Schmidlin P. Radiographic evaluation of different techniques for ridge preservation after tooth extraction: a randomized controlled clinical trial. J Clin Periodontol. 2013 Jan;40(1):90-8. doi: 10.1111/jcpe.12027. Epub 2012 Nov 19. PMID 23163915
- [Background] Chappuis V, Bornstein MM, Buser D, Belser U. Influence of implant neck design on facial bone crest dimensions in the esthetic zone analyzed by cone beam CT: a comparative study with a 5-to-9-year follow-up. Clin Oral Implants Res. 2016 Sep;27(9):1055-64. doi: 10.1111/clr.12692. Epub 2015 Sep 15. PMID 26370904
- [Background] Schropp L, Wenzel A, Spin-Neto R, Stavropoulos A. Fate of the buccal bone at implants placed early, delayed, or late after tooth extraction analyzed by cone beam CT: 10-year results from a randomized, controlled, clinical study. Clin Oral Implants Res. 2015 May;26(5):492-500. doi: 10.1111/clr.12424. Epub 2014 Jun 2. PMID 24890861